CLINICAL TRIAL: NCT00562458
Title: ARIMIDEX Study ( Non-interventional Study to Evaluate Arimidex in Adjuvant Therapy in Partial or Complete Response or Stabilized Disease After First Line Chemotherapy in Postmenopausal Women With Advanced Breast Cancer)
Brief Title: Non-interventional Study to Evaluate Arimidex in Postmenopausal Women With Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ARO-HCH-2006/1
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced breast cancer; Advanced breast cancer in postmenopausal women
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anastrozole

SUMMARY:
To evaluate Arimidex 6 month therapy as an adjuvant treatment in postmenopausal patients with advanced breast cancer in whom a partial or complete response or stabilized disease were obtained with first line chemotherapy, by tumoral response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be included in the program are that ones according to the indications specified in the Romanian anastrozole (Arimidex) approved SmPC (attached to the protocol)and who are already treated with anastrozole for at least 1 month before inclusion in this program/non-interventional study.

Exclusion Criteria:

* Patients not to be included in the programme: patients who have a known hypersensitivity to anastrozole (Arimidex®) or any of its excipients.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal patients with advanced breast cancer in whom a partial or complete response or stabilized disease were obtained with first line chemotherapy, by tumoral response assessment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-12